CLINICAL TRIAL: NCT02106546
Title: Randomized, Double-Blind, Multicenter, Phase 3 Study Comparing Veliparib Plus Carboplatin and Paclitaxel Versus Placebo Plus Carboplatin and Paclitaxel in Previously Untreated Advanced or Metastatic Squamous Non-Small Cell Lung Cancer (NSCLC)
Brief Title: Study Comparing Veliparib Plus Carboplatin and Paclitaxel Versus Placebo Plus Carboplatin and Paclitaxel in Previously Untreated Advanced or Metastatic Squamous Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M11-089; 2013-005020-42 (EudraCT Number)
Expanded Access: NCT03123211 (No longer available)
Record Dates: First submitted 2014-04-04; First posted 2014-04-08 (Estimated); Last update posted 2020-11-17 (Actual); Status verified 2020-10

CONDITIONS: Squamous Non-Small Cell Lung Cancer
Keywords: veliparib; carboplatin; paclitaxel; Poly Adenosine diphosphate (ADP)-ribose Polymerase (PARP); Overall Survival; Advanced; Metastatic; ABT-888; Squamous; Randomized; non-small cell lung cancer; placebo controlled
MeSH Terms: conditions — Neoplasm Metastasis; Carcinoma, Non-Small-Cell Lung | interventions — Carboplatin; veliparib; Paclitaxel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | US Export: No

ARMS (2):
- Veliparib + Carboplatin + Paclitaxel (Experimental): Participants received veliparib 120 mg orally twice daily (BID) on Days -2 to 5 (7 consecutive days) of each 21-day cycle and carboplatin at an area under the concentration-time curve (AUC) 6 mg/mL/min and paclitaxel 200 mg/m² by intravenous (IV) infusion on Day 1 of each 21-day cycle for up to a maximum 6 cycles of treatment, until treatment toxicity which, in the Investigator's opinion, prohibited further therapy, or until radiographic progression.
  Interventions: Drug: Carboplatin; Drug: Veliparib; Drug: Paclitaxel
- Placebo + Carboplatin + Paclitaxel (Placebo Comparator): Participants received placebo orally BID on Days -2 to 5 (7 consecutive days) of each 21-day cycle and carboplatin at an AUC 6 mg/mL/min and paclitaxel 200 mg/m² by IV infusion on Day 1 of each 21-day cycle for up to a maximum 6 cycles of treatment, until treatment toxicity which, in the Investigator's opinion, prohibited further therapy, or until radiographic progression.
  Interventions: Drug: Carboplatin; Drug: Paclitaxel; Drug: Placebo to veliparib

INTERVENTIONS:
Drug: Carboplatin — Carboplatin administered intravenously over approximately 15 to 30 minutes at (AUC 6 mg/mL/min) immediately following paclitaxel infusion.
Drug: Veliparib — Capsules taken orally twice a day, 12 hours apart.
  Other Names: ABT-888
  Arms: Veliparib + Carboplatin + Paclitaxel
Drug: Paclitaxel — Paclitaxel administered intravenously over 3 hours at a dose of 200 mg/m².
Drug: Placebo to veliparib — Capsules taken orally twice a day, 12 hours apart.
  Arms: Placebo + Carboplatin + Paclitaxel

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of the addition of veliparib plus carboplatin and paclitaxel versus the addition of placebo plus carboplatin and paclitaxel in adults with advanced or metastatic squamous non-small cell lung cancer (NSCLC).

ELIGIBILITY:
Inclusion Criteria:

1. Life expectancy > 12 weeks
2. Subject must have cytologically or histologically confirmed squamous NSCLC.
3. Subject must have advanced or metastatic squamous NSCLC that is not amenable to surgical resection or radiation with curative intent at time of study Screening.
4. Subjects with recurrent squamous NSCLC after surgical treatment that is not amenable to surgical resection or radiation with curative intent are eligible.
5. Subject must have at least 1 unidimensional measurable NSCLC lesion on a computerized tomography (CT) scan as defined by Response Evaluation Criteria In Solid Tumors (RECIST - version 1.1).

Exclusion Criteria:

1. Subject has a known hypersensitivity to paclitaxel or to other drugs formulated with polyethoxylated castor oil (Cremophor).
2. Subject has a known hypersensitivity to platinum compounds.
3. Subject has peripheral neuropathy >= grade 2.
4. Subject has non-squamous NSCLC, or a known epidermal growth factor receptor (EGFR) mutation of exon 19 deletion or L858R mutation in exon 21, or a known anaplastic lymphoma kinase (ALK) gene rearrangement.
5. Subject has received prior cytotoxic chemotherapy (including definitive chemoradiotherapy) for NSCLC, except for adjuvant or neoadjuvant therapy.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 970 (Actual)
Dates: Start 2014-04-10 (Actual); Primary Completion 2017-01-03 (Actual); Study Completion 2019-11-20 (Actual)

PRIMARY OUTCOMES:
Overall Survival (OS) in current smokers | Up to 3 years from first dose of study drug
  Time to death for a given subject will be defined as the number of days from the date that the subject was randomized to the date of the subject's death.

SECONDARY OUTCOMES:
Overall Survival (OS) in all subjects | Up to 3 years from first dose of study drug
  Time to death for a given subject will be defined as the number of days from the date that the subject was randomized to the date of the subject's death.
Progressive-Free Survival (PFS) in current smokers and in all subjects | Up to 3 years from first dose of study drug
  Defined as the number of days from the date that the subject was randomized to the date the subject experiences an event of disease progression or to the date of death (all causes of mortality) if disease progression is not reached.
Objective Response Rate (ORR) in current smokers and in all subjects | Up to 3 years from first dose of study drug
  Objective response rate is defined as the proportion of subjects with complete or partial response as determined by the investigator per RECIST (version 1.1)

OTHER OUTCOMES:
Change in Quality of Life: European Organisation for Research and Treatment of Cancer Quality of Life Core 30 Question Questionnaire (EORTC-QLQ-C30). | From Screening (prior to dosing) up to 2 years
Change in Quality of Life: European Organisation for Research and Treatment of Cancer Quality of Life Lung Cancer 13 Question Questionnaire (EORTC-LC13). | From Screening (prior to dosing) up to 2 years
Change in Eastern Cooperative Oncology Group (ECOG) Performance Status | From Screening (prior to dosing) up to 2 years
Change in Quality of Life: European Quality of Life-5 Dimensions-5 Levels Questionnaire (EQ-5D-5L) | From Screening (prior to dosing) up to 2 years
Duration of Response | From complete or partial response to disease progression (up to 3 years from randomization).
  The duration of overall response for a given subject will be defined as the number of days from the day the criteria are met for Complete or Partial Response (whichever is recorded first) to the date that Progressive Disease (PD) is objectively documented.

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie
Locations (225):
- United States (38):
  - Northeast Arkansas Clinical Ch /ID# 128071, Jonesboro, Arkansas
  - LA Hem-Oncology Med Group /ID# 129178, Los Angeles, California
  - VA Eastern Colorado Healthcare System /ID# 128065, Aurora, Colorado
  - Holy Cross Hospital /ID# 128074, Fort Lauderdale, Florida
  - University of Florida - Archer /ID# 126476, Gainesville, Florida
  - Cancer Specialists of North Florida - Southpoint /ID# 127815, Jacksonville, Florida
  - Winship Cancer Institute of Emory University /ID# 124061, Atlanta, Georgia
  - St. Luke's Mountain States Tumor Institute - Boise /ID# 124059, Boise, Idaho
  - Illinois Cancer Specialists /ID# 127468, Arlington Heights, Illinois
  - NorthShore University HealthSystem - Evanston Hospital /ID# 128585, Evanston, Illinois
  - Ingalls Memorial Hosp /ID# 128360, Harvey, Illinois
  - Midwestern Regional CTC /ID# 126124, Zion, Illinois
  - Goshen Center for Cancer Care /ID# 123875, Goshen, Indiana
  - Franciscan St. Francis Health /ID# 126678, Indianapolis, Indiana
  - Appalachian Regional Healthcare, Inc (ARH) /ID# 128061, Hazard, Kentucky
  - Henry Ford Health System /ID# 126500, Detroit, Michigan
  - Sparrow Regional Cancer Center, Sparrow Health System /ID# 127156, Lansing, Michigan
  - Minnesota Oncology Hematology, PA /ID# 127473, Minneapolis, Minnesota
  - Nebraska Hematology Oncology /ID# 127699, Lincoln, Nebraska
  - SE Nebraska Hema/Oncology Consultants P.C.d/b/a Southeast Nebraska Cancer Center /ID# 126477, Lincoln, Nebraska
  - Comprehensive Cancer Ctrs Neva /ID# 127491, Las Vegas, Nevada
  - Dartmouth-Hitchcock Medical Center /ID# 128075, Lebanon, New Hampshire
  - Hackensack Univ Med Ctr /ID# 124057, Hackensack, New Jersey
  - Gabrail Cancer Center Research /ID# 127415, Canton, Ohio
  - Penn State University and Milton S. Hershey Medical Center /ID# 126676, Hershey, Pennsylvania
  - The Jones Clinic, PC /ID# 124062, Germantown, Tennessee
  - Texas Oncology - Austin Midtown /ID# 127477, Austin, Texas
  - Texas Oncology - South Austin /ID# 127476, Austin, Texas
  - Parkland Health and Hosp Syste /ID# 128518, Dallas, Texas
  - Texas Oncology- Baylor Charles A. Sammons Cancer Center /ID# 128385, Dallas, Texas
  - UT Southwestern Medical Center /ID# 127876, Dallas, Texas
  - University of Texas MD Anderson Cancer Center /ID# 127946, Houston, Texas
  - Texas Oncology - Paris /ID# 127484, Paris, Texas
  - Texas Oncology - Waco /ID# 127459, Waco, Texas
  - University of Vermont Medical Center /ID# 128064, Burlington, Vermont
  - Virginia Oncology Associates /ID# 127458, Norfolk, Virginia
  - Northwest Cancer Specialists, P.C. /ID# 127486, Vancouver, Washington
  - Northwest Cancer Specialists, P.C. /ID# 127488, Vancouver, Washington
- Australia (6):
  - Southern Medical Day Care Ctr /ID# 125604, Wollongong, New South Wales
  - Sunshine Coast University Hosp /ID# 125608, Birtinya, Queensland
  - The Townsville Hospital /ID# 125609, Douglas, Queensland
  - Flinders Centre for Innovation /ID# 125605, Bedford Park, South Australia
  - The Queen Elizabeth Hospital /ID# 125607, Woodville, South Australia
  - Barwon Health University Hospital Geelong /ID# 125606, Geelong, Victoria
- Ordensklinikum Linz GmbH, Elisabethinen /ID# 126183, Linz, Austria
- Belarus (5):
  - Bobruysk Interdistrict Onco. /ID# 128999, Babruysk
  - Brest Regional Hospital /ID# 125955, Brest
  - State Institution Republican Scientific Practical Center of Oncology and Medica /ID# 125815, Lesnoy
  - Mogilev Reg Clin Oncology Dis /ID# 128639, Mogilev
  - Vitebsk Reg Clin Onc Disp /ID# 125516, Vitebsk
- Brazil (6):
  - Hospital Sao Lucas da PUCRS /ID# 127737, Porto Alegre, Rio Grande do Sul
  - Clinica de Neoplasias Litoral - Centro de Novos Tratamentos Itajai /ID# 127738, Itajaí, Santa Catarina
  - Fundacao Pio XII - Hospital de Cancer de Barretos /ID# 126736, Barretos, São Paulo
  - Instituto Nacional de Câncer José de Alencar Gomes da Silva (INCA) /ID# 127309, Rio de Janeiro
  - Instituto COI de Educacao e Pesquisa /ID# 127739, Rio de Janeiro
  - Fundacao Antonio Prudente - AC Camargo Cancer Center /ID# 126737, São Paulo
- Canada (9):
  - University of Calgary /Id# 126326, Calgary, Alberta
  - Cross Cancer Institute /ID# 126154, Edmonton, Alberta
  - Juravinski Cancer Clinic /ID# 126153, Hamilton, Ontario
  - Victoria Hospital /ID# 126669, London, Ontario
  - The Ottawa Hospital /ID# 126522, Ottawa, Ontario
  - Princess Margaret Cancer Centre /ID# 126155, Toronto, Ontario
  - McGill Univ HC /ID# 130431, Montreal, Quebec
  - Iucpq-Ul /Id# 126524, Québec, Quebec
  - CSSS Alphonse-Desjardins, CHAU de Levis /ID# 126149, Québec, Quebec
- Croatia (4):
  - Klinika za plucne bolesti Jordanovac /ID# 126537, Zagreb, City of Zagreb
  - Klinicki bolnicki centar Osijek /ID# 132214, Osijek, County of Osijek-Baranja
  - Opca bolnica Pula /ID# 126540, Pula
  - Opca bolnica Dr. Josip Bencevi /ID# 126539, Slavonski Brod
- Czechia (5):
  - Fakultni Nemocnice Olomouc /ID# 125820, Olomouc, Olomoucký kraj
  - Nemocnice Na Plesi s.r.o. /ID# 125817, Nová Ves pod Pleší, Pribram
  - Nemocnice Kyjov, prispevkova organizace /ID# 125819, Kyjov
  - Nemocnice Novy Jicin /ID# 125818, Nový Jičín
  - Vitkovicka nemocnice a. s. /ID# 127023, Ostrava
- Denmark (2):
  - Herlev Hospital /ID# 125995, Herlev, Capital Region
  - Odense Universitets Hospital /ID# 125996, Odense C, Region Syddanmark
- Egypt (4):
  - University of Alexandria /ID# 128337, Alexandria
  - Naser Institute for Res & Dev /ID# 129263, Cairo
  - Cairo Uni Hosp Al Kasr El Ainy /ID# 128338, Cairo
  - Cairo Uni Hosp Al Kasr El Ainy /ID# 128340, Cairo
- Estonia (2):
  - North Estonian Medical Centre /ID# 128215, Tallinn
  - Tartu University Hospital /ID# 127735, Tartu
- Finland (2):
  - Helsinki Univ Central Hospital /ID# 125897, Helsinki
  - Vaasa Central Hospital /ID# 125896, Vaasa
- France (9):
  - CHU Hopital Nord /ID# 128388, Marseille, Bouches-du-Rhone
  - Hopital Haut-Lévêque /ID# 135270, Pessac, Gironde
  - CHRU Lille - Hôpital Claude Huriez /ID# 126353, Lille, Hauts-de-France
  - Centre Hospitalier Le Mans /ID# 127902, Le Mans, Sarthe
  - Centre Hosp Intercommunal de Creteil /ID# 125922, Créteil, Val-de-Marne
  - CHRU de Brest - Hopital Morvan /ID# 127903, Brest
  - Centre Antoine Lacassagne /ID# 126360, Nice
  - Hospital Pontchaillou /ID# 126356, Rennes
  - Hopital Larrey - CHU de Toulouse /ID# 128394, Toulouse
- Germany (5):
  - Charite-Univ. Berlin, Benjamin-Franklin /ID# 125708, Berlin
  - Lungen Clinic Grosshansdorf /ID# 126107, Großhansdorf
  - Klinikum Kassel /ID# 127025, Kassel
  - Klinik Loewenstein GmbH /ID# 126191, Löwenstein
  - Univ Johannes Gutenberg /ID# 125603, Mainz
- Greece (4):
  - Papageorgiou General Hospital Thessaloniki /ID# 125876, Nea Efkarpia, Thessaloniki
  - General Hospital of Chest Diseases of Athens SOTIRIA /ID# 125879, Athens
  - Metropolitan Hospital /ID# 125878, Athens
  - University General Hospital of Heraklion PA.G.N.I /ID# 125877, Heraklion
- Hungary (10):
  - CRU Hungary Egeszsegugyi és Szolgaltato Kft. /ID# 135234, Miskolc, Borsod-Abauj Zemplen county
  - Orszagos Koranyi Pulmonologiai Intezet /ID# 126112, Budapest XII, Budapest
  - Debreceni Egyetem Klinikai Központ /ID# 126119, Debrecen
  - Veszprem Megyei Tudogyogyintez /ID# 126121, Farkasgyepű
  - Petz Aladar Megyei Oktato Korh /ID# 126110, Győr
  - Bekes Megyei Pandy Kalman Korhaz /ID# 126117, Gyula
  - Matrahaza Gyogyintezet /ID# 126109, Kékesteto
  - Fejer Megyei Szent Gyorgy Korh /ID# 126118, Székesfehérvár
  - Jasz-Nagykun-Szolnok Megyei Hetenyi Geza Korhaz /ID# 126120, Szolnok
  - Tudogyogyintezet Toeroekbalint /ID# 126111, Törökbálint
- Ireland (5):
  - St. James's Hospital /ID# 126177, Dublin, Dublin
  - Cork University Hospital /ID# 126176, Cork
  - Beaumont Hospital /ID# 126218, Dublin
  - University Hospital Limerick /ID# 126175, Limerick
  - University Hospital Waterford /ID# 126178, Waterford
- Israel (4):
  - Assaf Harofeh Medical Center /ID# 127076, Be’er Ya‘aqov
  - Hadassah University Hospital /ID# 127077, Jerusalem
  - Meir Medical Center /ID# 127078, Kfar Saba
  - Sheba Medical Center /ID# 127079, Ramat Gan
- Italy (7):
  - AO San Giuseppe Moscati /ID# 125701, Avellino
  - Istituto Europeo di Oncologia /ID# 125702, Milan
  - Azienda Ospedaliera San Gerardo di Monza _ Oncologia Medica /ID# 125704, Monza
  - A.O.U. San Luigi Gonzaga /ID# 125700, Orbassano
  - Azienda Ospedaliero Uni Parma /ID# 125703, Parma
  - Azienda Ospedaliera-Universitaria di Perugia-Divisione di Oncologia Medica. /ID# 125699, Perugia
  - Istituto Oncologico del Medite /ID# 132844, Viagrande
- Latvia (2):
  - Riga East Clinical Univ Hosp /ID# 125597, Riga
  - P. Stradins Clinical Univ Hosp /ID# 126322, Riga
- Lithuania (2):
  - Hospital of Lithuanian University of Health Sciences Kaunas Clinics /ID# 127176, Kaunas, Kaunas County
  - National Cancer Institute /ID# 126323, Vilnius
- Mexico (3):
  - Centro Estatal de Cancerologia /ID# 127583, Chihuahua City
  - Cancerologia de Queretaro S.C. /ID# 125920, Querétaro City
  - Hospital Angeles Centro Medico /ID# 127620, San Luis Potosí City
- Netherlands (7):
  - Jeroen Bosch Ziekenhuis /ID# 125709, 's-Hertogenbosch
  - Vrije Universiteit Medisch Centrum /ID# 125578, Amsterdam
  - Amphia Ziekenhuis /ID# 126466, Breda
  - Catharina Ziekenhuis /ID# 125577, Eindhoven
  - Ziekenhuis St. Jansdal /ID# 125576, Harderwijk
  - Atrium-Orbis Zuyderland Medisch Centrum /ID# 125710, Heerlen
  - Isala /ID# 125579, Zwolle
- Wellington Hospital (Capital and Coast District Health Board) /ID# 125755, Wellington, New Zealand
- Norway (6):
  - Haukeland University Hospital /ID# 126338, Bergen, Hordaland
  - Nordland Hospital /ID# 126337, Bodø
  - Sorlandet Sykehus HF /ID# 126341, Kristiansand
  - Oslo Universitetssykehus, Radiumhospitalet /ID# 126335, Oslo
  - Stavanger University Hospital /ID# 126336, Stavanger
  - Sykehuset i Vestfold HF /ID# 126340, Tønsberg
- Poland (4):
  - Mrukmed. Lekarz Beata Madej Mruk i Partner /ID# 126548, Rzeszów, Podkarpackie Voivodeship
  - Szpital Morski im. PCK /ID# 126547, Gdynia
  - NZOZ Magodent Ctr. Med. Ostro /ID# 126545, Warsaw
  - Mazowiecki Szpital Onkologiczn /ID# 126546, Wieliszew
- Portugal (6):
  - Hospital Senhora da Oliveira de Guimaraes, EPE /ID# 126761, Guimarães, Braga District
  - CCA Braga - Hospital de Braga /ID# 125837, Braga
  - Ctr Hosp Univ Coimbra, EPE /ID# 125838, Coimbra
  - Hospital Pulido Valente /ID# 125835, Lisbon
  - IPO Porto FG, EPE /ID# 125836, Porto
  - Centro Hospitalar de Sao Joao, EPE /ID# 125875, Porto
- VA Caribbean Healthcare System /ID# 124562, San Juan, Puerto Rico
- Russia (10):
  - Federal State Budgetary Scientific Institution N.N. Blokhin Russian Cancer Resea /ID# 128458, Moscow, Moscow
  - Sverdlovsk Regional Oncology Center Dispensary /ID# 128457, Yekaterinburg, Sverdlovsk Oblast
  - Volgograd Regional Clinical Oncology Dispensary /ID# 126350, Volgograd, Volgograd Oblast
  - Belgorod Oncology Dispensary /ID# 129899, Belgorod
  - State Budgetary Healthcare Institution"Irkutsk Regional Oncology Center /ID# 128460, Irkutsk
  - State Regional Budgetary Healthcare Institution " Murmansk Regional Oncology Dis /ID# 128461, Murmansk
  - Orenburg Regional Clinical Onc /ID# 137474, Orenburg
  - Ogarev Mordovia State Univ /ID# 127595, Saransk
  - Smolensk Regional Onc Clin Dis /ID# 127144, Smolensk
  - Cancer Research Institute Siberian Branch of the Russian Academy of Medical Scie /ID# 127143, Tomsk
- Serbia (5):
  - Clinical Center Serbia /ID# 128738, Belgrade, Beograd
  - Clinical Center of Nis /ID# 128735, Niš, Nisavski Okrug
  - Institute for Oncology and Rad /ID# 128721, Belgrade
  - University Hospital Bezanijska /ID# 128761, Belgrade
  - Institute For Pulmonary Diseas /ID# 128737, Kamenitz
- Slovakia (2):
  - Univerzitna Nemocnica Bratislava /ID# 126342, Bratislava
  - MEDEON, s.r.o. /ID# 128517, Pieštany
- South Africa (9):
  - GVI Oncology /ID# 126102, Port Elizabeth, Eastern Cape
  - Wits Clinical Research Site /ID# 126101, Johannesburg, Gauteng
  - Sandton Oncology Centre /ID# 126097, Johannesburg, Gauteng
  - University of Pretoria /ID# 127297, Pretoria, Gauteng
  - Dr Albert, Bouwer and Jordaan Incorporated /ID# 126098, Pretoria, Gauteng
  - Mary Potter Oncology Centre /ID# 126099, Pretoria, Gauteng
  - The Oncology Centre /ID# 126096, Durban, KwaZulu-Natal
  - Netcare Oncology Intervent Ctr /ID# 126100, Cape Town, Western Cape
  - Cancercare Outeniqua Oncology Unit /ID# 126103, George, Western Cape
- Spain (6):
  - Hospital Duran i Reynals /ID# 125161, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitario Puerta de Hierro Majadahonda /ID# 125160, Majadahonda, Madrid
  - Hospital Universitario Vall d'Hebron /ID# 125159, Barcelona
  - Hospital Universitario HM Sanchinarro /ID# 125162, Madrid
  - Hospital Universitario Virgen del Rocio /ID# 125207, Seville
  - Fundacion Instituto Valenciano Oncologia IVO /ID# 125205, Valencia
- Sweden (4):
  - Gavle Sjukhus /ID# 126444, Gävle
  - Sahlgrenska University Hosp /ID# 129997, Gothenburg
  - University Hospital Linkoping /ID# 126443, Linköping
  - Karolinska Univ Sjukhuset /ID# 126445, Solna
- Switzerland (4):
  - Kantonsspital St. Gallen /ID# 126349, Sankt Gallen, Canton of St. Gallen
  - Hirslanden Medical Center /ID# 128216, Aarau
  - Inselspital, Universitaetsklinik /ID# 126347, Bern
  - Spital STS AG /ID# 126348, Thun
- Turkey (Türkiye) (5):
  - Akdeniz University Medical Fac /ID# 126997, Antalya
  - Istanbul University-Cerrahpasa, Cerrahpasa Medical Faculty /ID# 126186, Istanbul
  - Marmara University Medical Fac /ID# 126187, Istanbul
  - Ege University Medical Faculty /ID# 126189, Izmir
  - Dr. Suat Seren Gogus Has /ID# 126190, Izmir
- Ukraine (7):
  - Communal non-profit enterprise Regional Center of Oncology /ID# 128221, Kharkiv, Kharkivs’ka Oblast’
  - Cherkassy Regional Onc Ctr /ID# 128222, Cherkasy
  - Regional Municipal Non-Profit Enterprise Bukovynian Clinical Oncology Center /ID# 128220, Chernivtsi
  - Municipal Non-Profit Enterprise City Clinical Hospital No.4 of Dnipro City Counc /ID# 128217, Dnipro
  - Lviv Oncological Regional Therapeutical and Diagnostic Centre /ID# 128218, Lviv
  - Poltava Regional Clinical Oncology Centre of Poltava Regional Council /ID# 128223, Poltava
  - Municipal Non-Profit Enterprise of Sumy Regional Council Sumy Regional Clinical /ID# 128219, Sumy
- United Kingdom (13):
  - Cheltenham General Hospital /ID# 125692, Cheltenham, Gloucestershire
  - Guy's and St Thomas' NHS Found /ID# 125694, London, London, City of
  - Norfolk and Norwich Univ Hosp /ID# 125697, Norwich, Norfolk
  - Betsi Cadwaladr Univ Health Bo /ID# 127177, Bangor
  - North Devon District Hospital /ID# 125689, Barnstaple
  - The Royal Bournemouth Hospital /ID# 125690, Bournemouth
  - East Kent Hosp Univ NHS Trust /ID# 125698, Canterbury
  - Gartnavel General Hospital /ID# 126233, Glasgow
  - James Paget University Hosp /ID# 125696, Great Yarmouth
  - Charing Cross Hospital /ID# 125688, London
  - Maidstone Hospital /ID# 125693, Maidstone
  - The Clatterbridge Cancer Ctr /ID# 125695, Metropolitan Borough of Wirral
  - The Newcastle Upon Tyne Hospitals NHS Foundation Trust Freeman Hospital /ID# 129228, Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols and clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data requests can be submitted at any time and the data will be accessible for 12 months, with possible extensions considered.
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous, independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA). For more information on the process, or to submit a request, visit the following link.
URL: https://www.abbvie.com/our-science/clinical-trials/clinical-trials-data-and-information-sharing/data-and-information-sharing-with-qualified-researchers.html

REFERENCES:
- [Derived] Ramalingam SS, Novello S, Guclu SZ, Bentsion D, Zvirbule Z, Szilasi M, Bernabe R, Syrigos K, Byers LA, Clingan P, Bar J, Vokes EE, Govindan R, Dunbar M, Ansell P, He L, Huang X, Sehgal V, Glasgow J, Bach BA, Mazieres J. Veliparib in Combination With Platinum-Based Chemotherapy for First-Line Treatment of Advanced Squamous Cell Lung Cancer: A Randomized, Multicenter Phase III Study. J Clin Oncol. 2021 Nov 10;39(32):3633-3644. doi: 10.1200/JCO.20.03318. Epub 2021 Aug 26. PMID 34436928